CLINICAL TRIAL: NCT03779347
Title: Prospective, Observational Study to Assess the Performance of CAA Measurement as a Diagnostic Tool for the Detection of Schistosoma Haematobium Infections in Pregnant Women and Their Newborn and Child in Lambaréné, Gabon
Brief Title: Schistosomiasis Diagnosis Using a CAA Antigen Test
Acronym: FreebiLyGAB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Principal Investigator, Prof. Ayola Akim ADEGNIKA, Director, Centre de Recherche Médicale de Lambaréné
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: FreebiLyGAB
Record Dates: First submitted 2018-12-08; First posted 2018-12-19 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Schistosomiasis Hematobium; Diagnostic; Drug Reaction; Pregnancy
Keywords: pregnancy, UPC-LF CAA, Schistosomiasis, children
MeSH Terms: conditions — Disease; Drug-Related Side Effects and Adverse Reactions; Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study assessor /investigator will be blinded from the treatment allocation. Treatment for study participants will be given under the supervision of the trained nurses at the ANC, while the study assessor will assess participants for clinical events at the research center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Schistosomiasis treated during pregnancy (Experimental): Praziquantel 40mg/kg once will be given during pregnancy at second to third trimester
  Interventions: Drug: Praziquantel
- Schistosomiasis treated after pregnancy (Active Comparator): Praziquantel 40mg/kg once will be given to parturient after delivery during lactation
  Interventions: Drug: Praziquantel
- All study participants (Experimental): UCP-LF CAA and composite diagnostic reference test based on extensive egg microscopy, plus serology, plus qPCR on egg DNA, and plus POC-CC will be used to detect schistosomiasis infection in pregnant women
  Interventions: Diagnostic Test: UCP-LF CAA; Diagnostic Test: composite diagnostic

INTERVENTIONS:
Drug: Praziquantel — Praziquantel to treat schistosomiasis during pregnancy
  Other Names: PZQ
  Arms: Schistosomiasis treated after pregnancy; Schistosomiasis treated during pregnancy
Diagnostic Test: UCP-LF CAA — UCP-LF CAA to diagnose Schistosomiasis during pregnancy
  Other Names: CAA
  Arms: All study participants
Diagnostic Test: composite diagnostic — composite diagnostic reference test based on extensive egg microscopy, serology, qPCR on egg DNA, and POC-CCA to diagnose Schistosomiasis during pregnancy
  Other Names: Composite
  Arms: All study participants

SUMMARY:
Schistosomiasis is one of most important human parasitic diseases worldwide. Pregnant women and their infants are two vulnerable population groups, particularly in sub-Saharan Africa, where - amongst other infectious agents - they are heavily exposed to infections with S. haematobium. Adoption of the recommendation and implementation by national disease control programs was however delayed in most African countries, due to the lack of safety data in humans and in the unborn babies. First results from randomized controlled trials with PZQ in pregnant women meanwhile have provided evidence for the safety of PZQ also in newborns.

In Gabon, S. haematobium is the primarily prevalent Schistosoma species infection. As it is true for most of observational and interventional studies on schistosomiasis, the power of the study is weakened due to the low sensitivity of reference schistosomiasis diagnosis applied, and one might correctly assume that a considerable proportion of samples were misclassified as negative in the control groups. Therefore, diagnostic tests that are highly sensitive and specific are essential to the detection of Schistosoma infections and are urgently needed for a test-and-treat strategy to control schistosomiasis in pregnancy as well as tools to determine efficacy of new interventions tested in clinical trials. Circulating anodic antigen (CAA) and circulating cathodic antigen (CCA) have levels correlating with the number of worms and have also been shown to clear within a few days or weeks after successful treatment. Assays measuring serum levels of these antigens (POC-CCA, UCP-LF CAA) are therefore deemed to assess drug efficacy.

Based on above mentioned tools, we decided to assess the accuracy of CAA measurement to determine the Schistosoma infection in two specific conditions: A) as a diagnostic tool for S. haematobium to prepare for the future implementation of a PZQ test-and-treat strategy and B) as a diagnostic tool to measure efficacy of praziquantel in schistosomiasis and pregnancy intervention trials.

DETAILED DESCRIPTION:
Study design

The freeBILy-GAB study is a set of interlinked prospective, observational studies conducted in Gabon to comprehensively assess the performance of CAA measurement for the detection of S. haematobium infections in pregnant women and infants. The study is composed of 3 sub-studies each targeted to assess a specific objective (see figure 1 for a schematic trial design, procedures and stages). The study activities will also contribute to safety reporting of PZQ use in pregnant women.

Sub-study A: At baseline, a diagnostic study will be conducted that will also allow to select sub-study B study participants. The approach is a prospective, cross-sectional, observational study conducted in pregnant women to determine the sensitivity and specificity of the UCP-LF CAA test for the detection of S. haematobium infections using urine samples. In the absence of a sensitive reference standard test, the index test (UCP-LF CAA) will be compared against a composite diagnostic reference test based on extensive egg microscopy, serology, qPCR on egg DNA, and POC-CCA. Sampling will include standardized urine collection of 3 consecutive days for S. haematobium diagnosis by egg microscopy, UCP-LF CAA testing, qPCR, and POC-CCA, one (1) stool sample (within the 3 days of urine sampling) to control for S. intercalatum and soil-transmitted helminths infections, and 1 blood sample (within the 3 days of urine sampling) to measure anti-Schistosoma antibodies and to detect any other parasitic infections endemic in the region including filarial and Plasmodia spps. and to provide blood cell counts and hemoglobin to assess pregnant women health status. The laboratory staff involved in performing the laboratory assays using the new techniques will be trained prior to the start of the study. Volunteers positive for any parasitic infection except filaria will be treated for the respective parasitic infection (S. haematobium, STH and malaria parasites) following national treatment guidelines. Women positive for S. haematobium by egg microscopy or UCP-LF CAA at baseline will receive either PZQ treatment (1x 40 mg/kg) within 7 days after the third urine sample (early PZQ treatment) or after delivery (late PZQ treatment) following an allocation ratio of 3:1. The late PZQ treatment group serves as a safety control group of PZQ administration to pregnant women and exposure of their offspring (s). Maternal and perinatal safety and efficacy outcomes will be assessed. For efficacy in offspring, birthweight (with low birthweight defined as weight at birth <2.5 kg) and small gestational age (used as an indicator for possible intrauterine growth restriction) will be investigated. In addition, the exposure to PZQ during pregnancy will be evaluated in infants at the age of 12 and 24 months. For efficacy in mothers, maternal anemia (defined as Hb < 11 g/dl) at inclusion and at delivery will be investigated.

Sub-study B is an observational, follow-up study of pregnant women infected with S. haematobium by egg microscopy and/or UCP-LF CAA test and treated with PZQ or intended for late PZQ treatment (see sub-study A). The aim of this sub-study is to assess if the UCP-LF CAA test can be used to evaluate treatment efficacy of PZQ during pregnancy. Women positive for S. haematobium by egg microscopy and/or UCP-LF CAA test and treated with PZQ (see sub-study A) will be actively followed-up. Urine will be collected on day 2, day 4 and day 6 after PZQ treatment to determine the kinetics of CAA decay and then once a week until both egg microscopy as well UCP-LF CAA assay become negative but no longer than 6 weeks after PZQ treatment.

Sub-study C is an observational, longitudinal study on mothers and their newborn babies. This sub-study aims to determine the incidence of S. haematobium infections and age to first S. haematobium infection in life time in infants born from mothers included in the study. Therefore, between 6 and 24 months post-delivery, mother and her infant will be asked to provide urine every three month until UCP-LF CAA test becomes positive for S. haematobium detection. In addition a questionnaire addressing water contact of mother and infant will be applied. If UCP-LF CAA test becomes positive, mothers will be treated with 1x 40 mg/kg PZQ.

Furthermore, outcome of PZQ treatment during pregnancy on infant development will be assessed at the age of 12 and 24 months after delivery in the two groups (early and late PZQ treatment groups). This allows for a comparison to the freeBILy-MAD study in Madagascar.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational age comprised between 16 and 30 weeks (based on last date of menses)
* Willing to deliver in one of the four maternities: three in Lambaréné and one in Fougamou
* Provide a written informed consent for both themselves and for newborn follow-up or the written informed consent by the legal guardian if pregnant woman is a minor

Exclusion Criteria:

* - Willing to move out of the study area within the coming 24 months
* Known having a medically confirmed complicated pregnancy a complicated pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
UPC-LF CAA performance | first two years of the study
  Test performance of the UCP-LF CAA test for the detection of S. haematobium infection in pregnancy (sub-study A)
Egg reduction rate | first two years of the study
  Egg reduction rate after PZQ treatment (sub-study B)
CAA reduction rate | first two years of the study
  CAA reduction and after PZQ treatment (sub-study B)
Prevalence of S. hematobium in children using UCP-LF CAA | last two years of the study
  Prevalence of S. haematobium infections in infants below two years of age in our study areas as determined by UCP-LF CAA test (sub-study C)
Prevalence of S. hematobium in children using microscopy | last two years of the study
  Prevalence of S. haematobium infections in infants below two years of age in our study areas as determined by egg microscopy

SECONDARY OUTCOMES:
Clinical safety assessment upon PZQ intake | anytime after drug administration until the last born child reach two years old.
  Adverse events related and or unrelated to PZQ administration to pregnant women will be assessed clinically:
  * During pregnancy
  * At delivery
  * During the first two years of unborn child
Efficacy rate using microscopy | first two years of the study
  PZQ Cure rate for S. haematobium treatment in pregnancy (sub-study B) assessed by microscopy test
Efficacy rate using UCP-LF CAA test | first two years of the study
  PZQ Cure rate for S. haematobium treatment in pregnancy (sub-study B) assessed by UCP-LF CAA test

CONTACTS AND LOCATIONS:
Overall Officials: Ayola A ADEGNIKA, MD, PhD, Principal Investigator — Centre de Recherches Médicales de Lambaréné (CERMEL); Andrea Kreidenweiss, PhD, Study Chair — University Hospital Tuebingen
Locations (2):
- Gabon (2):
  - Centre de Recherches Médicales de Lambaréné, Lambaréné, Moyen-Ogooué Province
  - Centre de Recherches Medicales de Lambaréné, Lambaréné

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Honkpehedji YJ, Adegnika AA, Dejon-Agobe JC, Zinsou JF, Mba RB, Gerstenberg J, Rakotozandrindrainy R, Rakotoarivelo RA, Rasamoelina T, Sicuri E, Schwarz NG, Corstjens PLAM, Hoekstra PT, van Dam GJ, Kreidenweiss A; freeBILy Consortium. Prospective, observational study to assess the performance of CAA measurement as a diagnostic tool for the detection of Schistosoma haematobium infections in pregnant women and their child in Lambarene, Gabon: study protocol of the freeBILy clinical trial in Gabon. BMC Infect Dis. 2020 Sep 29;20(1):718. doi: 10.1186/s12879-020-05445-1. PMID 32993559